CLINICAL TRIAL: NCT02310503
Title: Spanish Registry of Mohs Surgery [Registro Español de Cirugía de Mohs]
Brief Title: Spanish Registry of Mohs Surgery
Acronym: REGESMOHS
Status: Completed | Type: Observational
Sponsor: Fundación Academia Española de Dermatología (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: FAE-MOH-2013-01
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Dermatofibrosarcoma; Melanoma; Histiocytoma, Malignant Fibrous; Neoplasms, Adnexal and Skin Appendage
Keywords: Mohs Surgery
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Dermatofibrosarcoma; Melanoma; Histiocytoma, Malignant Fibrous; Neoplasms, Adnexal and Skin Appendage | interventions — Mohs Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mohs surgery: Patients treated using Mohs surgery. Other exposures considered include patient characteristics, preoperative care and technical variants.
  Interventions: Procedure: Mohs surgery

INTERVENTIONS:
Procedure: Mohs surgery — A surgical technique used primarily in the treatment of skin neoplasms, especially basal cell or squamous cell carcinoma of the skin. This procedure is a microscopically controlled excision of cutaneous tumors either after fixation in vivo or after freezing the tissue. Serial examinations of fresh tissue specimens are most frequently done.

SUMMARY:
REGESMOHS (Registro Español de cirugía de Mohs) aims at describing effectiveness of Mohs surgery, and patient, tumor and technique factors related to adverse events and tumor recurrence.

REGESMOHS is a prospective cohort, including all patients considered for Mohs surgery in participating centers. All consecutive patients are included. The only exclusion criteria are being under 18-years-old or legally incompetent. Pre-planned follow-up is as required by common clinical practice, but at least once a year for the study period.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients considered for Mohs surgery

Exclusion Criteria:

* Under 18 years-old
* Legally incompetent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients considered for Mohs surgery in participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2013-07-01; Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Tumor recurrence | 6 years

SECONDARY OUTCOMES:
Short term outcomes | 1 month
  Bleeding, infection, abnormal scar, necrosis
Use of resources | During surgery
  Need for admission, type of anesthesia, number of surgical steps, participating doctors,time in surgery room.
Impairments of body function and structure | 6 years
  presence of: abnormal scar, ectropion, nostril alteration, oral sphincter incompetence,other

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garcia-Doval, MD, PhD, Study Director — Research Unit. Academia Española de Dermatologia y Venereologia (Spanish Academy of Dermatology)
Locations (15):
- Spain (15):
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital del Mar, Barcelona
  - Hospital Quirón Teknon, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Complejo Hospitalario Universitario de Guadalajara, Guadalajara
  - Complejo Asistencial Universitario de León, León
  - Clínica Quirón, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital La Zarzuela, Madrid
  - Hospital Universitario Fundación de Alcorcón, Madrid
  - Clínica Universitaria de Navarra, Pamplona
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Manises, Valencia
  - Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso-Alonso T, Redondo-Bellon P, Sanmartin-Jimenez O, de Eusebio-Murillo E, Garcia-Doval I, Rodriguez-Prieto MA. Census of Centers That Perform Mohs' Micrographic Surgery in Spain and Description of Their Activity: A Feasibility Study for the Mohs' Micrographic Surgery Registry of the Foundation of the Spanish Academy of Dermatology and Venereology. Actas Dermosifiliogr. 2015 Nov;106(9):764-6. doi: 10.1016/j.ad.2015.02.014. Epub 2015 Jun 23. No abstract available. English, Spanish. PMID 26115794
- [Background] Ruiz-Salas V, Garces JR, Minano Medrano R, Alonso-Alonso T, Rodriguez-Prieto MA, Lopez-Estebaranz JL, Sanmartin-Jimenez O, Guillen Barona C, Delgado Jimenez Y, Toll-Abello A, Vargas Diez E, Ciudad Blanco C, Alfaro Rubio A, Allende Markixana I, de Eusebio Murillo E, Manubens-Mercade E, Vazquez-Veiga H, Barchino Ortiz L, Garcia-Doval I, Redondo Bellon P. Description of Patients Undergoing Mohs Surgery in Spain: Initial Report on Data From the Spanish Registry of Mohs Surgery (REGESMOHS). Actas Dermosifiliogr. 2015 Sep;106(7):562-8. doi: 10.1016/j.ad.2015.04.002. Epub 2015 May 28. English, Spanish. PMID 26028578
- [Background] de Eusebio Murillo E, Martin Fuentes A, Ruiz-Salas V, Garces JR, Minano Medrano R, Lopez-Estebaranz JL, Alonso-Alonso T, Rodriguez-Prieto MA, Delgado Jimenez Y, Morales V, Redondo Bellon P, Manubens-Mercade E, Sanmartin-Jimenez O, Guillen Barona C, Cabeza R, Cano N, Toll-Abello A, Navarro Tejedor R, Artola Igarza JL, Allende Markixana I, Alfaro Rubio A, Ciudad Blanco C, Vazquez-Veiga H, Barchino Ortiz L, Descalzo MA, Garcia-Doval I. Characterization of Surgical Procedures in the Spanish Mohs Surgery Registry (REGESMOHS) for 2013-2015. Actas Dermosifiliogr. 2017 Nov;108(9):836-843. doi: 10.1016/j.ad.2017.04.018. Epub 2017 Aug 9. English, Spanish. PMID 28802488
- [Background] Camarero-Mulas C, Delgado Jimenez Y, Sanmartin-Jimenez O, Garces JR, Rodriguez-Prieto MA, Alonso-Alonso T, Minano Medrano R, Lopez-Estebaranz JL, de Eusebio Murillo E, Redondo P, Ciudad-Blanco C, Toll-Abello A, Artola Igarza JL, Allende Markixana I, Suarez Fernandez R, Alfaro Rubio A, Alonso Pacheco ML, Vazquez-Veiga H, de la Cueva Dobao P, Ruiz-Salas V, Vilarrasa Rull E, Barchino L, Morales-Gordillo V, Ocerin-Guerra I, Navarro Tejedor R, Hueso L, Mayor Arenal M, Seoane-Pose MJ, Cano-Martinez N, Garcia-Doval I, Descalzo MA; REGESMOHS (Registro Espanol de Cirugia de Mohs). Mohs micrographic surgery in the elderly: comparison of tumours, surgery and first-year follow-up in patients younger and older than 80 years old in REGESMOHS. J Eur Acad Dermatol Venereol. 2018 Jan;32(1):108-112. doi: 10.1111/jdv.14586. Epub 2017 Oct 5. PMID 28898467
- [Background] Ruiz-Salas V, Garces JR, Alonso-Alonso T, Rodriguez-Prieto MA, Toll-Abello A, Eusebio Murillo E, Minano R, Lopez-Estebaranz JL, Sanmartin-Jimenez O, Guillen Barona C, Allende Markixana I, Alfaro Rubio A, Delgado Jimenez Y, Navarro R, Barchino Ortiz L, Lazaro Ochaita P, Vilarasa E, Ciudad Blanco C, Vazquez-Veiga H, Artola Igarza JL, Alonso ML, Garcia-Doval I, Descalzo MA, Redondo Bellon P. Description of patients excluded for Mohs surgery after pre-surgical evaluation: data from the Regesmohs Spanish registry. Actas Dermosifiliogr (Engl Ed). 2018 May;109(4):346-350. doi: 10.1016/j.ad.2017.11.008. Epub 2018 Jan 17. English, Spanish. PMID 29373111
- [Background] Delgado Jimenez Y, Camarero-Mulas C, Sanmartin-Jimenez O, Garces JR, Rodriguez-Prieto MA, Alonso-Alonso T, Minano Medrano R, Lopez-Estebaranz JL, de Eusebio Murillo E, Redondo P, Ciudad-Blanco C, Toll A, Artola Igarza JL, Allende Markixana I, Suarez Fernandez R, Alfaro Rubio A, Alonso Pacheco ML, Vazquez-Veiga H, de la Cueva Dobao P, Ruiz-Salas V, Vilarrasa E, Barchino L, Morales-Gordillo V, Ocerin-Guerra I, Navarro Tejedor R, Hueso L, Mayor Arenal M, Seoane-Pose MJ, Cano-Martinez N, Garcia-Doval I, Descalzo MA; REGESMOHS. Differences of Mohs micrographic surgery in basal cell carcinoma versus squamous cell carcinoma. Int J Dermatol. 2018 Nov;57(11):1375-1381. doi: 10.1111/ijd.14223. Epub 2018 Sep 23. PMID 30246444
- See also: Updated descrition of the study (in Spanish) — https://aedv.es/investigacion/proyectos-de-investigacion/registro-nacional-de-cirugia-micrografica-de-mohs/